CLINICAL TRIAL: NCT07129122
Title: A Novel Technique for Percutaneous Mitral Paravalvular Leak Closure: LBBAP Lead Assisted Ventricular Septal Way
Status: Completed | Type: Observational
Sponsor: Bursa Postgraduate Hospital (Other)
Responsible Party: Principal Investigator, Hasan ARI, Professor Doctor, Bursa Postgraduate Hospital
Other Study IDs: Bursa YIEAH Case
Record Dates: First submitted 2025-08-02; First posted 2025-08-19 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Mitral Paravalvular Leaks (PVL)

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Transventricular access: Paravalvular leak
  Interventions: Other: Transventricular access

INTERVENTIONS:
Other: Transventricular access — Transventricular access will perform with LBBAP lead from left subclavian way.

SUMMARY:
The investigators will perform closure the mitral paravalvular leak in patient with mechanical aortic and mitral valve.

DETAILED DESCRIPTION:
The mitral mitral paravalvular leak closure access are left atrial and transapical in patient with mechanical aortic and mitral valve.

In this case the investigators will use interventricular septal access.

ELIGIBILITY:
Inclusion Criteria:

* Had mitral paravalvüler leak Had mitral and aortic mechanical valve

Exclusion Criteria:

* Not suitable for left subclavian access Active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with prosthetic mitral valve and paravalvular leakage
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2025-07-31 (Actual); Primary Completion 2025-08-02 (Actual); Study Completion 2025-08-02 (Actual)

PRIMARY OUTCOMES:
mitral paravalvüler leak closure sucsess | 2 day

OTHER OUTCOMES:
mitral paravalvüler leak closure sucsess without complication | 2 day

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Yüksek İhtisas Eğitim ve Araştırma Hastanesi, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No